CLINICAL TRIAL: NCT01371747
Title: A Multicenter, Randomized, Open-Label, Dose Ranging Study to Evaluate the Efficacy and Safety of Patiromer in the Treatment of Hyperkalemia in Patients With Hypertension and Diabetic Nephropathy Receiving Angiotensin-converting Enzyme Inhibitor (ACEI) and/or Angiotensin II Receptor Blocker (ARB) Drugs, With or Without Spironolactone
Brief Title: Patiromer in the Treatment of Hyperkalemia in Patients With Hypertension and Diabetic Nephropathy (AMETHYST-DN)
Acronym: AMETHYST-DN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Relypsa, Inc. (Industry)
Responsible Party: Sponsor
Organization: Vifor Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RLY5016-205; 2011-000165-12 (EudraCT Number)
Record Dates: First submitted 2011-06-09; First posted 2011-06-13 (Estimated); Results first posted 2015-12-17 (Estimated); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Chronic Kidney Disease; Hypertension; Hyperkalemia
Keywords: Hyperkalemia; Chronic Kidney Disease; Treatment of Hyperkalemia; Hypertension; Diabetic Nephropathy
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension; Hyperkalemia; Diabetic Nephropathies | interventions — patiromer; Suspensions; Losartan; Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Stratum 1: 8.4 g/d patiromer (Experimental): Participants with baseline serum potassium > 5.0 to 5.5 mEq/L (milliequivalent)
  Interventions: Drug: patiromer; Drug: losartan; Drug: spironolactone
- Stratum 1: 16.8 g/d patiromer (Experimental): Participants with baseline serum potassium > 5.0 to 5.5 mEq/L
  Interventions: Drug: patiromer; Drug: losartan; Drug: spironolactone
- Stratum 1: 25.2 g/d patiromer (Experimental): Participants with baseline serum potassium > 5.0 to 5.5 mEq/L
  Interventions: Drug: patiromer; Drug: losartan; Drug: spironolactone
- Stratum 2: 16.8 g/d patiromer (Experimental): Participants with baseline serum potassium > 5.5 to < 6.0 mEq/L
  Interventions: Drug: patiromer; Drug: losartan; Drug: spironolactone
- Stratum 2: 25.2 g/d patiromer (Experimental): Participants with baseline serum potassium > 5.5 to < 6.0 mEq/L
  Interventions: Drug: patiromer; Drug: losartan; Drug: spironolactone
- Stratum 2: 33.6 g/d patiromer (Experimental): Participants with baseline serum potassium > 5.5 to < 6.0 mEq/L
  Interventions: Drug: patiromer; Drug: losartan; Drug: spironolactone

INTERVENTIONS:
Drug: patiromer — Cohorts 1, 2 and 3 - Patiromer starting dose: 8.4 g/day, orally, as a divided dose, twice daily. The dose of patiromer could be titrated based on participant's serum potassium response (Stratum 1)
  Other Names: RLY5016 for Oral Suspension; Veltassa
  Arms: Stratum 1: 8.4 g/d patiromer
Drug: patiromer — Cohorts 1, 2 and 3 - Patiromer starting dose: 16.8 g/day, orally, as a divided dose, twice daily. The dose of patiromer could be titrated based on participant's serum potassium response. (Stratum 2)
  Other Names: RLY5016 for Oral Suspension; Veltassa
  Arms: Stratum 2: 16.8 g/d patiromer
Drug: patiromer — Cohorts 1, 2 and 3 - Patiromer starting dose: 16.8 g/day, orally, as a divided dose, twice daily. The dose of patiromer could be titrated based on participant's serum potassium response (Stratum 1)
  Other Names: RLY5016 for Oral Suspension; Veltassa
  Arms: Stratum 1: 16.8 g/d patiromer
Drug: patiromer — Cohorts 1, 2 and 3 - Patiromer starting dose: 25.2 g/day, orally, as a divided dose, twice daily. The dose of patiromer could be titrated based on participant's serum potassium response (Stratum 1)
  Other Names: RLY5016 for Oral Suspension; Veltassa
  Arms: Stratum 1: 25.2 g/d patiromer
Drug: patiromer — Cohorts 1, 2 and 3 - Patiromer starting dose: 25.2 g/day, orally, as a divided dose, twice daily. The dose of patiromer could be titrated based on participant's serum potassium response. (Stratum 2)
  Other Names: RLY5016 for Oral Suspension; Veltassa
  Arms: Stratum 2: 25.2 g/d patiromer
Drug: patiromer — Cohorts 1, 2 and 3 - Patiromer starting dose: 33.6 g/day, orally, as a divided dose, twice daily. The dose of patiromer could be titrated based on participant's serum potassium response. (Stratum 2)
  Other Names: RLY5016 for Oral Suspension; Veltassa
  Arms: Stratum 2: 33.6 g/d patiromer
Drug: losartan — losartan dose: 100 mg/d, oral, once daily (initiated during Run-In Period; Cohort 1)
Drug: spironolactone — Spironolactone dose: 25 mg/d or up to 50 mg/d, oral, once daily (initiated during Run-In Period; Cohort 2)

SUMMARY:
This study determined the optimal starting dose of patiromer in treating hyperkalemia in participants with hypertension and diabetic nephropathy who were already receiving ACEI and/or ARB drugs, with or without spironolactone. This study also evaluated the efficacy and safety of patiromer and the long term use of patiromer.

DETAILED DESCRIPTION:
RLY5016-205 was an open-label, randomized, dose ranging study to determine the optimal starting dose, efficacy and safety of patiromer in treating hyperkalemia in hypertensive patients with nephropathy due to type 2 diabetes mellitus (T2DM) who were already receiving Angiotensin-converting Enzyme Inhibitor (ACEI) and/or Angiotensin II Receptor Blocker (ARB) drugs, with or without spironolactone.

The study consisted of the following periods:

* Screening: Up to 10 days (1 visit)
* Run-in for those who were not hyperkalemic at screening (Cohorts 1 and 2): up to 4 weeks (1 to 4 visits)
* Patiromer Treatment Initiation: first 8 weeks of patiromer treatment (a minimum of 10 visits)
* Patiromer Long-Term Maintenance: additional 44 weeks of patiromer treatment up to a total of one year (minimum of 11 additional visits)
* Follow-up (after patiromer discontinuation): 1 week (2 visits) OR 4 weeks (5 visits) depending on the final serum potassium level

ELIGIBILITY:
Inclusion Criteria:

1. Age 30 - 80 years old at screening (S1)
2. Type 2 diabetes mellitus (T2DM) diagnosed after age 30 which has been treated with oral medications or insulin for at least 1 year prior to S1
3. Chronic kidney disease (CKD): estimated glomerular filtration rate (eGFR) 15 - < 60 mL/min/1.73m2 at screening based on central lab serum creatinine measurement (except for participants with hyperkalemia at S1), whose eligibility will be assessed based on local lab eGFR value)
4. Urine albumin/creatinine ratio (ACR):

   1. Cohorts 1 and 2: urine ACR ≥ 30 mg/g at S1 AND average urine ACR ≥ 30 mg/g at the beginning of Run-In Period (R0) based on up to three ACR values obtained starting at S1 and ending at the R0 Visit
   2. Cohort 3: not applicable
5. Local laboratory serum potassium (K+) values of:

   1. Cohorts 1 and 2: 4.3 - 5.0 mEq/L at S1; AND 4.5 - 5.0 mEq/L at R0; AND > 5.0 - < 6.0 mEq/L at randomization to patiromer (Baseline, T0 Visit)
   2. Cohort 3: > 5.0 - < 6.0 mEq/L at S1 OR at R0 after same day confirmation
6. Must be receiving an ACEI and/or ARB for at least 28 days prior to screening
7. Average systolic blood pressure (SBP) ≥ 130 - < 180 mmHg AND average DBP ≥ 80 - < 110 mmHg (sitting) at both screening and R0 (as applicable)
8. Females of child-bearing potential must be non-lactating, must have a negative serum pregnancy test at screening, and must have used a highly effective form of contraception for at least 3 months before patiromer administration, during the study, and for one month after study completion
9. Provide their written informed consent prior to participation in the study

Exclusion Criteria:

1. Type 1 diabetes mellitus
2. Central lab hemoglobin A1c > 12% at Screening 1 (S1) (except for Cohort 3 participants who are hyperkalemic at S1)
3. Emergency treatment for T2DM within the last 3 months
4. A confirmed SBP > 180 mmHg or diastolic blood pressure (DBP) > 110 mmHg at any time during SI or Run-In Period or at Baseline T0 Visit
5. Central lab serum magnesium < 1.4 mg/dL (< 0.58 mmol/L) at screening (Cohort 3 participants will be evaluated based on local lab serum magnesium measurement)
6. Central lab urine ACR ≥ 10000 mg/g at screening (except for Cohort 3 participants who are hyperkalemic at S1)
7. Confirmed diagnosis or history of renal artery stenosis (unilateral or bilateral)
8. Diabetic gastroparesis
9. Non-diabetic chronic kidney disease
10. History of bowel obstruction, swallowing disorders, severe gastrointestinal disorders or major gastrointestinal surgery (e.g., large bowel resection)
11. Current diagnosis of NYHA (New York Heart Association) Class III or IV heart failure
12. Body mass index (BMI) ≥ 40 kg/m2
13. Any of the following events having occurred within 2 months prior to screening: unstable angina as judged by the Principal Investigator (PI), unresolved acute coronary syndrome, cardiac arrest or clinically significant ventricular arrhythmias, transient ischemic attack or stroke, use of any intravenous cardiac medication
14. Prior kidney transplant, or anticipated need for transplant during study participation
15. Active cancer, currently on cancer treatment or history of cancer in the past 2 years except for non-melanocytic skin cancer which is considered cured
16. History of alcoholism or drug/chemical abuse within 1 year
17. Central lab liver enzymes [alanine aminotransferase (ALT), aspartate aminotransferase (AST)] > 3 times upper limit of normal at S1 (except for Cohort 3 patients with hyperkalemia at S1, who will have local lab ALT and AST)
18. Loop and thiazide diuretics or other antihypertensive medications (calcium channel blocker, beta-blocker, alpha-blocker, or centrally acting agent) that have not been stable for at least 28 days prior to screening or not anticipated to remain stable during study participation
19. Current use of polymer-based drugs (e.g., sevelamer, sodium polystyrene sulfonate, colesevelam, colestipol, cholestyramine), phosphate binders (e.g., lanthanum carbonate), or other potassium binders, or their anticipated need during study participation
20. Current use of lithium
21. Use of potassium sparing medications, including aldosterone antagonists (e.g., spironolactone), drospirenone, potassium supplements, bicarbonate or baking soda in the last 7 days prior to screening
22. Use of any investigational product within 30 days or 5 half-lives, whichever is longer, prior to screening
23. Inability to consume the investigational product, or, in the opinion of the Investigator, inability to comply with the protocol
24. In the opinion of the Investigator, any medical condition, uncontrolled systemic disease, or serious intercurrent illness that would significantly decrease study compliance or jeopardize the safety of the participant or affect the validity of the trial results

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2011-06; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director Clinical Operations, Study Director — Relypsa, Inc.
Locations (43):
- Croatia (6):
  - Investigator Site 201, Karlovac
  - Investigator Site 207, Osijek
  - Investigator Site 203, Rijeka
  - Investigator Site 202, Zagreb
  - Investigator Site 204, Zagreb
  - Investigator Site 208, Zagreb
- Georgia (11):
  - Investigator Site 305, Tbilisi
  - Investigator Site 309, Tbilisi
  - Investigator site 301, Tbilisi
  - Investigator Site 302, Tbilisi
  - Investigator Site 303, Tbilisi
  - Investigator Site 304, Tbilisi
  - Investigator Site 306, Tbilisi
  - Investigator Site 307, Tbilisi
  - Investigator Site 310, Tbilisi
  - Investigator Site 311, Tbilisi
  - Investigator Site 308, Tbilisi
- Hungary (14):
  - Investigator Site 508, Budapest
  - Investigator Site 502, Budapest
  - Investigator Site 514, Budapest
  - Investigator Site 513, Budapest
  - Investigator Site 517, Budapest
  - Investigator Site 522, Győr
  - Investigator Site 523, Hatvan
  - Investigator Site 515, Jászberény
  - Investigator Site 506, Kistarcsa
  - Investigator Site 503, Kisvárda
  - Investigator Site 510, Mosonmagyaróvár
  - Investigator Site 504, Székesfehérvár
  - Investigator Site 505, Szikszó
  - Investigator Site 507, Veszprém
- Serbia (6):
  - Investigator Site 601, Belgrade
  - Investigator Site 602, Belgrade
  - Investigator Site 604, Belgrade
  - Investigator Site 605, Belgrade
  - Investigator Site 603, Novi Sad
  - Investigator Site 607, Zrenjanin
- Slovenia (6):
  - Investigator Site 703, Celje
  - Investigator Site 706, Golnik
  - Investigator Site 708, Jesenice
  - Investigator Site 701, Maribor
  - Investigator Site 704, Slovenj Gradec
  - Investigator Site 707, Šempeter pri Gorici

REFERENCES:
- [Background] Bakris GL, Pitt B, Weir MR, Freeman MW, Mayo MR, Garza D, Stasiv Y, Zawadzki R, Berman L, Bushinsky DA; AMETHYST-DN Investigators. Effect of Patiromer on Serum Potassium Level in Patients With Hyperkalemia and Diabetic Kidney Disease: The AMETHYST-DN Randomized Clinical Trial. JAMA. 2015 Jul 14;314(2):151-61. doi: 10.1001/jama.2015.7446. PMID 26172895
- [Derived] Bakris GL, Woods SD, Alvarez PJ, Arthur SP, Kumar R. Hyperkalemia Management in Older Adults With Diabetic Kidney Disease Receiving Renin-Angiotensin-Aldosterone System Inhibitors: A Post Hoc Analysis of the AMETHYST-DN Clinical Trial. Kidney Med. 2021 Mar 13;3(3):360-367.e1. doi: 10.1016/j.xkme.2021.01.005. eCollection 2021 May-Jun. PMID 34136782
- [Derived] Natale P, Palmer SC, Ruospo M, Saglimbene VM, Strippoli GF. Potassium binders for chronic hyperkalaemia in people with chronic kidney disease. Cochrane Database Syst Rev. 2020 Jun 26;6(6):CD013165. doi: 10.1002/14651858.CD013165.pub2. PMID 32588430
- [Derived] Pitt B, Bakris GL, Weir MR, Freeman MW, Lainscak M, Mayo MR, Garza D, Zawadzki R, Berman L, Bushinsky DA. Long-term effects of patiromer for hyperkalaemia treatment in patients with mild heart failure and diabetic nephropathy on angiotensin-converting enzymes/angiotensin receptor blockers: results from AMETHYST-DN. ESC Heart Fail. 2018 Aug;5(4):592-602. doi: 10.1002/ehf2.12292. Epub 2018 May 16. PMID 29767459

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 324 participants were enrolled in the study; 306 participants were randomized to receive study drug.
Pre-assignment Details: Screening serum potassium ≤ 5 mEq/L (milliequivalent) entered Run-in: Cohort 1 stopped ACEI/ARB (angiotensin-converting enzyme inhibitor/angiotensin receptor blockers), started losartan; Cohort 2 started spironolactone; Run-in (Cohorts 1 and 2) or screening (Cohort 3) > 5 mEq/L entered study.
Groups:
- Stratum 1: 8.4 g/d Patiromer: Participants with baseline serum potassium > 5.0 - 5.5 mEq/L randomized to 8.4 g/day patiromer starting dose, orally, as a divided dose twice a day.
- Stratum 1: 16.8 g/d Patiromer: Participants with baseline serum potassium > 5.0 - 5.5 mEq/L randomized to 16.8 g/day patiromer starting dose, orally, as a divided dose twice a day.
- Stratum 1: 25.2 g/d Patiromer: Participants with baseline serum potassium > 5.0 - 5.5 mEq/L randomized to 25.2 g/day patiromer starting dose, orally, as a divided dose twice a day.
- Stratum 2: 16.8 g/d Patiromer: Participants with baseline serum potassium > 5.5 to < 6.0 mEq/L randomized to 16.8 g/day patiromer starting dose, orally, as a divided dose twice a day.
- Stratum 2: 25.2 g/d Patiromer: Participants with baseline serum potassium > 5.5 to < 6.0 mEq/L randomized to 25.2 g/day patiromer starting dose, orally, as a divided dose twice a day.
- Stratum 2: 33.6 g/d Patiromer: Participants with baseline serum potassium > 5.5 to < 6.0 mEq/L randomized to 33.6 g/day patiromer starting dose, orally, as a divided dose twice a day.
Period: Overall Study
Arm/Group | Stratum 1: 8.4 g/d Patiromer | Stratum 1: 16.8 g/d Patiromer | Stratum 1: 25.2 g/d Patiromer | Stratum 2: 16.8 g/d Patiromer | Stratum 2: 25.2 g/d Patiromer | Stratum 2: 33.6 g/d Patiromer
Started | 74 | 74 | 74 | 26 | 28 | 30
Completed | 56 | 51 | 50 | 17 | 21 | 16
Not Completed | 18 | 23 | 24 | 9 | 7 | 14
Not completed — Adverse Event | 4 | 2 | 7 | 2 | 2 | 2
Not completed — Death | 1 | 0 | 4 | 1 | 2 | 0
Not completed — Abnormal Renal Function | 0 | 2 | 0 | 1 | 0 | 1
Not completed — High Serum Potassium Results | 1 | 1 | 1 | 2 | 0 | 2
Not completed — Low Serum Potassium Results | 1 | 1 | 1 | 1 | 0 | 3
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Non-Compliance | 3 | 4 | 3 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 6 | 12 | 5 | 2 | 2 | 4
Not completed — Other Reasons | 2 | 1 | 2 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: 306 participants were randomized and stratified by baseline serum potassium (2 randomized participants in Stratum 1 did not receive any study drug: 1 participant withdrew consent and 1 participant was randomized in error and was withdrawn from the study); 304 participants were analyzed for safety.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum 1: 8.4 g/d Patiromer | Stratum 1: 16.8 g/d Patiromer | Stratum 1: 25.2 g/d Patiromer | Stratum 2: 16.8 g/d Patiromer | Stratum 2: 25.2 g/d Patiromer | Stratum 2: 33.6 g/d Patiromer | Total
Number analyzed (Participants) | 74 | 73 | 73 | 26 | 28 | 30 | 304
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 29 | 28 | 12 | 12 | 13 | 122
  >=65 years | 46 | 44 | 45 | 14 | 16 | 17 | 182
Age, Continuous [Median (Full Range); unit: years] | 67 [46 to 80] | 70 [37 to 79] | 68 [40 to 79] | 66.5 [56 to 76] | 68.5 [39 to 80] | 65 [44 to 78] | 67.5 [37 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 26 | 26 | 8 | 13 | 10 | 112
  Male | 45 | 47 | 47 | 18 | 15 | 20 | 192

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Change in Serum Potassium From Baseline to Week 4 or Time of First Titration for Each Individual Starting Dose Group
Description: Least square mean changes from Baseline to Week 4/first titration were derived from parallel lines ANCOVA model with randomized starting dose and baseline serum potassium value as covariates.
Time Frame: Baseline to Week 4 or First Titration which could occur at any scheduled study visit after patiromer initiation.
Population: Included all randomized participants who received at least 1 dose of patiromer. Analyses of endpoints included participants with available central laboratory potassium values at the time point of interest.
Measure: Least Squares Mean (Standard Error); unit: mEq/L
Arm/Group | Stratum 1: 8.4 g/d Patiromer | Stratum 1: 16.8 g/d Patiromer | Stratum 1: 25.2 g/d Patiromer | Stratum 2: 16.8 g/d Patiromer | Stratum 2: 25.2 g/d Patiromer | Stratum 2: 33.6 g/d Patiromer
Number analyzed (Participants) | 73 | 72 | 72 | 26 | 27 | 30
mEq/L | -0.35 (0.066) | -0.51 (0.067) | -0.55 (0.067) | -0.87 (0.134) | -0.97 (0.132) | -0.92 (0.125)
Statistical Analysis 1: Comparison: Stratum 1: 8.4 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value <0.001
Statistical Analysis 2: Comparison: Stratum 1: 16.8 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; p < 0.001, ANCOVA — P-Value <0.001
Statistical Analysis 3: Comparison: Stratum 1: 25.2 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value <0.001
Statistical Analysis 4: Comparison: Stratum 2: 16.8 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value <0.001
Statistical Analysis 5: Comparison: Stratum 2: 25.2 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value <0.001
Statistical Analysis 6: Comparison: Stratum 2: 33.6 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value <0.001

2. Secondary Outcome: Least Squares Mean Change in Serum Potassium From Baseline to Week 8 or Time of First Titration for Each Individual Starting Dose Group
Description: Least squares mean changes from Baseline to Week 8/first titration were derived from parallel lines ANCOVA model with randomized starting dose and baseline serum potassium value as covariates.
Time Frame: Baseline to Week 8 or First Titration which could occur at any scheduled study visit after patiromer initiation.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mEq/L
Arm/Group | Stratum 1: 8.4 g/d Patiromer | Stratum 1: 16.8 g/d Patiromer | Stratum 1: 25.2 g/d Patiromer | Stratum 2: 16.8 g/d Patiromer | Stratum 2: 25.2 g/d Patiromer | Stratum 2: 33.6 g/d Patiromer
Number analyzed (Participants) | 73 | 72 | 72 | 26 | 27 | 30
mEq/L | -0.35 (0.070) | -0.47 (0.070) | -0.54 (0.070) | -0.88 (0.142) | -0.95 (0.139) | -0.91 (0.132)
Statistical Analysis 1: Comparison: Stratum 1: 8.4 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; p < 0.001, ANCOVA — P-Value <0.001
Statistical Analysis 2: Comparison: Stratum 1: 16.8 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; p < 0.001, ANCOVA — P-Value <0.001
Statistical Analysis 3: Comparison: Stratum 1: 25.2 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value <0.001
Statistical Analysis 4: Comparison: Stratum 2: 16.8 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value <0.001
Statistical Analysis 5: Comparison: Stratum 2: 25.2 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value <0.001
Statistical Analysis 6: Comparison: Stratum 2: 33.6 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value <0.001

3. Secondary Outcome: Least Squares Mean Change in Serum Potassium From Baseline to Day 3 During the Treatment Initiation Period for Each Individual Starting Dose Group
Description: Least squares mean changes from Baseline to Day 3 were derived from parallel lines ANCOVA model with randomized starting dose and baseline serum potassium value as covariates.
Time Frame: Baseline to Day 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mEq/L
Arm/Group | Stratum 1: 8.4 g/d Patiromer | Stratum 1: 16.8 g/d Patiromer | Stratum 1: 25.2 g/d Patiromer | Stratum 2: 16.8 g/d Patiromer | Stratum 2: 25.2 g/d Patiromer | Stratum 2: 33.6 g/d Patiromer
Number analyzed (Participants) | 68 | 63 | 69 | 25 | 26 | 30
mEq/L | -0.26 (0.048) | -0.28 (0.050) | -0.31 (0.047) | -0.65 (0.086) | -0.59 (0.084) | -0.53 (0.079)
Statistical Analysis 1: Comparison: Stratum 1: 8.4 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; p < 0.001, ANCOVA — P-Value <0.001
Statistical Analysis 2: Comparison: Stratum 1: 16.8 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; p < 0.001, ANCOVA — P-Value <0.001
Statistical Analysis 3: Comparison: Stratum 1: 25.2 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value <0.001
Statistical Analysis 4: Comparison: Stratum 2: 16.8 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value <0.001
Statistical Analysis 5: Comparison: Stratum 2: 25.2 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value <0.001
Statistical Analysis 6: Comparison: Stratum 2: 33.6 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value <0.001

4. Secondary Outcome: Mean Change in Serum Potassium From Baseline to Week 52 During the Long-term Maintenance Period for Each Individual Starting Dose Group
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Stratum 1: 8.4 g/d Patiromer | Stratum 1: 16.8 g/d Patiromer | Stratum 1: 25.2 g/d Patiromer | Stratum 2: 16.8 g/d Patiromer | Stratum 2: 25.2 g/d Patiromer | Stratum 2: 33.6 g/d Patiromer
Number analyzed (Participants) | 50 | 49 | 44 | 15 | 19 | 15
mEq/L | -0.54 (0.465) | -0.44 (0.440) | -0.50 (0.417) | -1.00 (0.466) | -0.96 (0.414) | -1.17 (0.569)
Statistical Analysis 1: Comparison: Stratum 1: 8.4 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; Mean Difference (Net) = -0.54 — Estimated values were based on summary statistics
Statistical Analysis 2: Comparison: Stratum 1: 16.8 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; Mean Difference (Net) = -0.44 — Estimated values were based on summary statistics
Statistical Analysis 3: Comparison: Stratum 1: 25.2 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; Mean Difference (Net) = -0.50 — Estimated values were based on summary statistics
Statistical Analysis 4: Comparison: Stratum 2: 16.8 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; Mean Difference (Net) = -1.00 — Estimated values were based on summary statistics
Statistical Analysis 5: Comparison: Stratum 2: 25.2 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; Mean Difference (Net) = -0.96 — Estimated values were based on summary statistics
Statistical Analysis 6: Comparison: Stratum 2: 33.6 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; Mean Difference (Net) = -1.17 — Estimated values were based on summary statistics

5. Secondary Outcome: Mean Change in Serum Potassium From Week 52 or Last Patiromer Dose (if Occurred Before Week 52) to Follow-up Visits Plus 7 Days
Time Frame: Week 52 or Last Patiromer Dose (if Occurred before Week 52) to Following up Visit Plus 7 Days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Stratum 1: 8.4 g/d Patiromer | Stratum 1: 16.8 g/d Patiromer | Stratum 1: 25.2 g/d Patiromer | Stratum 2: 16.8 g/d Patiromer | Stratum 2: 25.2 g/d Patiromer | Stratum 2: 33.6 g/d Patiromer
Number analyzed (Participants) | 52 | 52 | 50 | 20 | 17 | 20
mEq/L | 0.36 (0.567) | 0.22 (0.424) | 0.30 (0.508) | 0.41 (0.660) | 0.39 (0.331) | 0.58 (0.557)
Statistical Analysis 1: Comparison: Stratum 1: 8.4 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; Mean Difference (Net) = 0.36 — Estimated values were based on summary statistics
Statistical Analysis 2: Comparison: Stratum 1: 16.8 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; Mean Difference (Net) = 0.22 — Estimated values were based on summary statistics
Statistical Analysis 3: Comparison: Stratum 1: 25.2 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; Mean Difference (Net) = 0.30 — Estimated values were based on summary statistics
Statistical Analysis 4: Comparison: Stratum 2: 16.8 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; Mean Difference (Net) = 0.41 — Estimated values were based on summary statistics
Statistical Analysis 5: Comparison: Stratum 2: 25.2 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; Mean Difference (Net) = 0.39 — Estimated values were based on summary statistics
Statistical Analysis 6: Comparison: Stratum 2: 33.6 g/d Patiromer; Each starting dose group was compared to its baseline; Test type: Superiority or Other; Mean Difference (Net) = 0.58 — Estimated values were based on summary statistics

6. Secondary Outcome: Proportion of Participants Achieving Serum Potassium Levels Within 3.5 to 5.5 mEq/L at Week 8 for Each Individual Starting Dose Group
Time Frame: Baseline to Week 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stratum 1: 8.4 g/d Patiromer | Stratum 1: 16.8 g/d Patiromer | Stratum 1: 25.2 g/d Patiromer | Stratum 2: 16.8 g/d Patiromer | Stratum 2: 25.2 g/d Patiromer | Stratum 2: 33.6 g/d Patiromer
Number analyzed (Participants) | 63 | 65 | 64 | 24 | 24 | 22
percentage of participants | 100 [94.3 to 100.0] | 100 [94.5 to 100] | 98.4 [91.6 to 100] | 91.7 [73.0 to 99.0] | 95.8 [78.9 to 99.9] | 95.5 [77.2 to 99.9]
Statistical Analysis 1: Comparison: Stratum 1: 8.4 g/d Patiromer; Test type: Superiority or Other; Percentage of Participants = 100, 95% CI 2-sided [94.3 to 100.0] — 2-sided 95% exact binomial CI
Statistical Analysis 2: Comparison: Stratum 1: 16.8 g/d Patiromer; Test type: Superiority or Other; Percentage of Participants = 100, 95% CI 2-sided [94.5 to 100] — 2-sided 95% exact binomial CI
Statistical Analysis 3: Comparison: Stratum 1: 25.2 g/d Patiromer; Test type: Superiority or Other; Percentage of Participants = 98.4, 95% CI 2-sided [91.6 to 100] — 2-sided 95% exact binomial CI
Statistical Analysis 4: Comparison: Stratum 2: 16.8 g/d Patiromer; Test type: Superiority or Other; Percentage of Participants = 91.7, 95% CI 2-sided [73 to 99] — 2-sided 95% exact binomial CI
Statistical Analysis 5: Comparison: Stratum 2: 25.2 g/d Patiromer; Test type: Superiority or Other; Percentage of Participants = 95.8, 95% CI 2-sided [78.9 to 99.9] — 2-sided 95% exact binomial CI
Statistical Analysis 6: Comparison: Stratum 2: 33.6 g/d Patiromer; Test type: Superiority or Other; Percentage of Participants = 95.5, 95% CI 2-sided [77.2 to 99.9] — 2-sided 95% exact binomial CI

7. Secondary Outcome: Proportion of Participants Achieving Serum Potassium Levels Within 4.0 to 5.0 mEq/L at Week 8 for Each Individual Starting Dose Group
Time Frame: Baseline to Week 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stratum 1: 8.4 g/d Patiromer | Stratum 1: 16.8 g/d Patiromer | Stratum 1: 25.2 g/d Patiromer | Stratum 2: 16.8 g/d Patiromer | Stratum 2: 25.2 g/d Patiromer | Stratum 2: 33.6 g/d Patiromer
Number analyzed (Participants) | 63 | 65 | 64 | 24 | 24 | 22
percentage of participants | 95.2 [86.7 to 99.0] | 90.8 [81.0 to 96.5] | 81.3 [69.5 to 89.9] | 79.2 [57.8 to 92.9] | 91.7 [73.0 to 99.0] | 77.3 [54.6 to 92.2]
Statistical Analysis 1: Comparison: Stratum 1: 8.4 g/d Patiromer; Test type: Superiority or Other; Percentage of Participants = 95.2, 95% CI 2-sided [86.7 to 99.0] — 2-sided 95% exact binomial CI
Statistical Analysis 2: Comparison: Stratum 1: 16.8 g/d Patiromer; Test type: Superiority or Other; Percentage of Participants = 90.8, 95% CI 2-sided [81.0 to 96.5] — 2-sided 95% exact binomial CI
Statistical Analysis 3: Comparison: Stratum 1: 25.2 g/d Patiromer; Test type: Superiority or Other; Percentage of Participants = 81.3, 95% CI 2-sided [69.5 to 89.9] — 2-sided 95% exact binomial CI
Statistical Analysis 4: Comparison: Stratum 2: 16.8 g/d Patiromer; Test type: Superiority or Other; Percentage of Participants = 79.2, 95% CI 2-sided [57.8 to 92.9] — 2-sided 95% exact binomial CI
Statistical Analysis 5: Comparison: Stratum 2: 25.2 g/d Patiromer; Test type: Superiority or Other; Percentage of Participants = 91.7, 95% CI 2-sided [73 to 99] — 2-sided 95% exact binomial CI
Statistical Analysis 6: Comparison: Stratum 2: 33.6 g/d Patiromer; Test type: Superiority or Other; Percentage of Participants = 77.3, 95% CI 2-sided [54.6 to 92.2] — 2-sided 95% exact binomial CI

8. Secondary Outcome: Time to First Serum Potassium Measurement of 4.0 - 5.0 mEq/L During Treatment Initiation Period for Each Individual Starting Dose Group
Time Frame: Baseline to Week 8
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Stratum 1: 8.4 g/d Patiromer | Stratum 1: 16.8 g/d Patiromer | Stratum 1: 25.2 g/d Patiromer | Stratum 2: 16.8 g/d Patiromer | Stratum 2: 25.2 g/d Patiromer | Stratum 2: 33.6 g/d Patiromer
Number analyzed (Participants) | 72 | 72 | 73 | 26 | 28 | 30
Days | 4 [4 to 5] | 4 [4 to 6] | 4 [4 to 5] | 8 [4 to 9] | 7.5 [4 to 8] | 8 [4 to 8]

9. Secondary Outcome: Proportions of Participants Achieving Serum Potassium Levels Within 3.8 to 5.0 mEq/L at Week 52 for Each Individual Starting Dose Group
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stratum 1: 8.4 g/d Patiromer | Stratum 1: 16.8 g/d Patiromer | Stratum 1: 25.2 g/d Patiromer | Stratum 2: 16.8 g/d Patiromer | Stratum 2: 25.2 g/d Patiromer | Stratum 2: 33.6 g/d Patiromer
Number analyzed (Participants) | 58 | 63 | 59 | 22 | 24 | 20
percentage of participants | 86.3 [73.7 to 94.3] | 81.6 [68.0 to 91.2] | 88.9 [75.9 to 96.3] | 86.7 [59.5 to 98.3] | 89.5 [66.9 to 98.7] | 93.3 [68.1 to 99.8]
Statistical Analysis 1: Comparison: Stratum 1: 8.4 g/d Patiromer; Test type: Superiority or Other; Percentage of Participants = 86.3, 95% CI 2-sided [73.7 to 94.3] — 2-sided 95% exact binomial CI
Statistical Analysis 2: Comparison: Stratum 1: 16.8 g/d Patiromer; Test type: Superiority or Other; Percentage of Participants = 81.6, 95% CI 2-sided [68.0 to 91.2] — 2-sided 95% exact binomial CI
Statistical Analysis 3: Comparison: Stratum 1: 25.2 g/d Patiromer; Test type: Superiority or Other; Percentage of Participants = 88.9, 95% CI 2-sided [75.9 to 96.3] — 2-sided 95% exact binomial CI
Statistical Analysis 4: Comparison: Stratum 2: 16.8 g/d Patiromer; Test type: Superiority or Other; Percentage of Participants = 86.7, 95% CI 2-sided [59.5 to 98.3] — 2-sided 95% exact binomial CI
Statistical Analysis 5: Comparison: Stratum 2: 25.2 g/d Patiromer; Test type: Superiority or Other; Percentage of Participants = 89.5, 95% CI 2-sided [66.9 to 98.7] — 2-sided 95% exact binomial CI
Statistical Analysis 6: Comparison: Stratum 2: 33.6 g/d Patiromer; Test type: Superiority or Other; Percentage of Participants = 93.3, 95% CI 2-sided [68.1 to 99.8] — 2-sided 95% exact binomial CI

ADVERSE EVENTS:
Time Frame: Up to 28 days after Week 52 or last patiromer dose, whichever was earlier
Description: Randomized participants who received at least one dose of trial medication
Arm/Group | Stratum 1: 8.4 g/d Patiromer | Stratum 1: 16.8 g/d Patiromer | Stratum 1: 25.2 g/d Patiromer | Stratum 2: 16.8 g/d Patiromer | Stratum 2: 25.2 g/d Patiromer | Stratum 2: 33.6 g/d Patiromer
Serious Adverse Events (participants affected / at risk) | 9/74 | 10/73 | 10/73 | 6/26 | 5/28 | 4/30
Other Adverse Events (participants affected / at risk) | 28/74 | 29/73 | 29/73 | 14/26 | 14/28 | 22/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum 1: 8.4 g/d Patiromer (N=74) | Stratum 1: 16.8 g/d Patiromer (N=73) | Stratum 1: 25.2 g/d Patiromer (N=73) | Stratum 2: 16.8 g/d Patiromer (N=26) | Stratum 2: 25.2 g/d Patiromer (N=28) | Stratum 2: 33.6 g/d Patiromer (N=30)
Acute left ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 0 | 1 | 0
Diabetic retinopathy (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Brain death (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sudden cardiac death (General disorders) | 0 | 0 | 3 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Arteriosclerotic gangrene (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Intraocular pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 1 | 1 | 2 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Nephropathy toxic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 2 | 1 | 1 | 1 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diabetic vascular disorder (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0
Femoral artery occlusion (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum 1: 8.4 g/d Patiromer (N=74) | Stratum 1: 16.8 g/d Patiromer (N=73) | Stratum 1: 25.2 g/d Patiromer (N=73) | Stratum 2: 16.8 g/d Patiromer (N=26) | Stratum 2: 25.2 g/d Patiromer (N=28) | Stratum 2: 33.6 g/d Patiromer (N=30)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 4 | 0 | 1 | 2
Angina pectoris (Cardiac disorders) | 0 | 1 | 2 | 1 | 2 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 1 | 2 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 2 | 4 | 2 | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 4 | 3 | 4 | 2 | 1 | 5
Diarrhoea (Gastrointestinal disorders) | 6 | 5 | 1 | 3 | 1 | 1
Influenza (Infections and infestations) | 3 | 0 | 4 | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 2 | 1 | 1 | 2
Urinary tract infection (Infections and infestations) | 3 | 3 | 2 | 0 | 2 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 2 | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 0 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 5 | 6 | 2 | 4 | 5
Headache (Nervous system disorders) | 3 | 2 | 1 | 0 | 0 | 2
Renal failure chronic (Renal and urinary disorders) | 5 | 4 | 2 | 2 | 3 | 6
Hypertension (Vascular disorders) | 5 | 7 | 2 | 4 | 2 | 4
Hypotension (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreements generally provide that PI cannot publish single site data before publication of the multi-site publication, unless 1 year has elapsed since completion of the study at all sites. Thereafter, PI may publish provided that PI shall: provide a copy of the publication to sponsor at least 60 days in advance of submission for publication; delete sponsor's confidential information as requested; and delay publication up to an additional 90 days to permit protection of intellectual property.